CLINICAL TRIAL: NCT04961411
Title: Colonic Gallstone Ileus: a Literature Review With a Diagnostic-therapeutic Algorithm
Brief Title: Colonic Gallstone Ileus, Diagnostic-therapeutic Algorithm
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tomislav Bruketa (Other)
Responsible Party: Sponsor-Investigator, Tomislav Bruketa, General and abdominaln surgeon, M.D., Ph.D., Clinical Hospital Centre Zagreb
Organization: Clinical Hospital Centre Zagreb (Other)
Other Study IDs: 01012021
Record Dates: First submitted 2021-06-25; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Gall Stone
Keywords: Gallstone ileus; Cholecystocolonic fistula; Risk factors; Diagnosis; Therapy; Algorithm
MeSH Terms: conditions — Gallstones; Disease | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- published cases of patients with gallstone ileus: We will observe clinical signs, diagnostic procedures and therapeutic procedures and options
  Interventions: Procedure: operation or non-operative treatment

INTERVENTIONS:
Procedure: operation or non-operative treatment — type of operation or if possible non-operative treatment

SUMMARY:
Gallstone ileus is a rare complication of gallstone disease. There is no systematic review on CGI. We analyze published literature on the subject and plan to propose a diagnostic-therapeutic algorithm for CGI. Following the Preferred Reporting Items for Systematic Reviews and Meta-Analysis (PRISMA) and AMSTAR (Assessing the methodological quality of systematic reviews) guidelines, we will performe a systematic review of English-, German-, Spanish-, Japanese-, and Italian-language articles using PubMed (1946-2021), PubMed Central (1900-2021), and Google Scholar.

The search items include 'gallstone ileus', 'colonic gallstone ileus', 'gallstone coleus', 'cholecystocolonic fistula', 'ileo biliar', 'iléus biliaire', 'ileo di calcoli biliary', 'galsteen ileus', 'fístula colecistocolônica', 'fistule cholécystocolique'. Additional studies will be identified by reviewing reference lists of retrieved studies. We will include all cases and case series with a complete description of CGI.

Exclusion criteria: (1) small bowel gallstone ileus; (2) gastric outlet gallstone ileus; (3) non-gallstone intraluminal obstruction; and (4) cholecystocolonic fistula without CGI.

The primary outcome: a relationship of demographic data, gallstone size, symptoms, obstruction level, risk factors, and comorbidities (biliary history, diverticular disease, cardiovascular disease, radiation of pelvis), diagnostics (palpable mass in the abdomen and rectal exam, laboratory tests, sigmoidoscopy/colonoscopy, x-ray, computed tomography (CT), colonic Rigler's triad) with the correct diagnosis.

The secondary outcome: the identification of therapeutic options and related survival.

The third outcome: to develop a comprehensive diagnostic-therapeutic algorithm for CGI.

The study is exempt from ethics approval because we synthesized data from published studies.

ELIGIBILITY:
Inclusion Criteria:

* all published cases and case series with a complete description of colonic gallstone ileus

Exclusion Criteria:

* small bowel gallstone ileus; gastric outlet gallstone ileus; non-gallstone intraluminal obstruction; and cholecystocolonic fistula without colonic gallstone ileus

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: We will take data from all accessible published case and case series with complete description of colonic gallstone ileus
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Demographic data | up to 8 weeks
  male to female ratio
Gallstone size | up to 8 weeks
  gallstone size
Symptoms | up to 8 weeks
  possible disease presentation
Obstruction level | up to 8 weeks
  level of obstruction in colon
Risk factors and comorbidities | up to 8 weeks
  biliary history, diverticular disease
Diagnostics - clinical exam | up to 8 weeks
  palpable mass in the abdomen
Diagnostics - endoscopy | up to 8 weeks
  Colonoscopy
Diagnostics - x-ray | up to 8 weeks
  plain abdominal x-ray
Diagnostics - computed tomography | up to 8 weeks
  Abdominal computed tomography
Diagnostics - specific signs | up to 8 weeks
  Colonic Rigler's triad

SECONDARY OUTCOMES:
Therapeutic options - operation without resection | up to 8 weeks
  number of patients with cololithotomy
Therapeutic options - operation with resection | up to 8 weeks
  number of patients with colonic resection
Therapeutic options - conservative treatment | up to 8 weeks
  number of patients treated conservatively
Survival | up to 8 weeks
  Survival of patients according to therapeutic option

CONTACTS AND LOCATIONS:
Overall Officials: Goran Augustin, M.D., Ph.D, Study Director — Clinical Hospital Centre Zagreb
Locations (1):
- University hospital center Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes
As a supplement data with publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: With publication with no time limit